CLINICAL TRIAL: NCT00537225
Title: Multifactor Risk Reduction for Optimal Management of PAD
Acronym: VIGOR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Stanford University (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OKR0001AGG/SGG
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; walking time; lifestyle modification; cardiovascular risk reduction; exercise; diet; claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity; Intermittent Claudication | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Home-based exercise
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-Exercise group (Experimental): Home based exercise
  Interventions: Behavioral: exercise
- B- Usual Care (No Intervention): Exercise as usually prescribed by provider

INTERVENTIONS:
Behavioral: exercise — tailored multifactor CVD risk reduction
  Arms: A-Exercise group

SUMMARY:
Patients with peripheral arterial disease (PAD) experience significant functional limitations due to ischemic symptoms (claudication) and are at high risk for CVD morbidity and mortality resulting from untreated cardiovascular disease (CVD) risk factors and aggressive atherosclerosis. The overall Goal of this randomized controlled clinical trial is to examine the synergistic effect of a multifactor risk reduction on walking distance, blood flow and quality of life in 300 patients with PAD.

Specifically, we will compare the effects of 24 months of a novel, yet well-tested multiple risk factor reduction program, the Health Education and Risk Reduction Training (HEAR2T) Program for PAD versus enhanced standard care on: 1) symptom limited walking distance as assessed by treadmill exercise testing and walking impairment questionnaire; 2) endothelial function as measured by flow mediated vasodilation (FMVD) via brachial artery ultrasound. We will also explore the association between FMVD and decreased oxidative stress (as measured by oxygen radical absorbance capacity and urinary isoprostanes) and reduced degradation of nitric oxide (NO) and/or increased NO biosynthesis (as measured by urine nitrogen oxide, plasma nitrogen oxide, plasma asymmetric dimethylarginine, plasma, urine and platelet cyclic GMP).

Secondary hypotheses examine the association between reducing CVD risk factors, improved endothelial function, increased walking distance, improved quality of life and number of metabolic syndrome abnormalities in PAD patients.

Significance. This study will contribute to evidence on the efficacy of multiple risk factor reduction on improving physical function and quality of life in the understudied, elderly PAD patient. This study will also provide preliminary evidence for the biological basis for the efficacy of multifactor risk reduction in restoring vascular homeostasis, critical because of its role in antiatherogenesis and maintaining vasoreactivity, both necessary for slowing the progression of atherosclerosis.

DETAILED DESCRIPTION:
closed to recruitment

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this study include:

1. Age 50 years or older with one or more CVD risk factor
2. PAD secondary to atherosclerosis with significant claudication
3. Claudication is defined as pain, ache, cramp, numbness or severe fatigue of muscles of one or both lower extremities, reproducibly provoked by walking causing the patient to slow or stop walking pace
4. Ankle-brachial index (ABI) < 0.90
5. In diabetics ABI is inaccurate, in which case, we will substitute toe pressures < 60 mmHg
6. ABI one minute after exercise is at least 20% lower than index leg resting ABI
7. Capable of walking at least 50 feet
8. Primary limitation to walking is claudication, not coexisting conditions such as severe CAD, uncontrolled hypertension, pulmonary disease, severe arthritis, or orthopedic conditions
9. Difference of walking time between two consecutive (of four) baseline treadmill tests must be < 25%.

Exclusion Criteria:

Exclusion criteria include:

1. Active malignancy or tumor or other condition that would severely limit life expectancy
2. Any type of major surgery during the last 3 months (i.e. aortic or lower extremity arterial surgery, angioplasty, or lumbar sympathectomy, leg amputation above the ankle)
3. Residence in a long-term institutional setting
4. Psychiatric disorders with currently active manifestations
5. Uncontrolled metabolic disorders (renal failure, liver failure, thyrotoxicosis)
6. Active symptoms suggestive of an acute coronary syndrome or decompensated heart failure
7. Lack of phone access (either by self or through neighbors/family members)
8. Other specified circumstances incompatible with case-management (i.e., plan to move away from area)
9. Presence of another household member or first-degree relative already enrolled in the study
10. Current enrollment in another clinical trial
11. Regular participation in an exercise program for at least 3 months prior to study entry.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
walking time | 24 months
  determined by symptom limited walking time on treadmill exercise test

SECONDARY OUTCOMES:
quality of life, biomarkers of CVD risk, endothelial function | 24 months
  Quality of life per SF-36; biomarkers include: lipids, endothelial function per FMD

CONTACTS AND LOCATIONS:
Overall Officials: Roberta K Oka, ANP, DNSc, Principal Investigator — PAIRE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oka RK, Conte MS, Owens CD, Rapp J, Fung G, Alley HF, Giacomini JC, Myers J, Mohler ER 3rd. Efficacy of optimal long-term management of multiple cardiovascular risk factors (CVD) on walking and quality of life in patients with peripheral artery disease (PAD): protocol for randomized controlled trial. Vasc Med. 2012 Feb;17(1):17-28. doi: 10.1177/1358863X11430886. PMID 22363015
- [Result] Oka RK, Alley HF. Differences in nutrition status by body mass index in patients with peripheral artery disease. J Vasc Nurs. 2012 Sep;30(3):77-87. doi: 10.1016/j.jvn.2012.04.003. PMID 22901446